CLINICAL TRIAL: NCT01499927
Title: Early Reassessment of Intravenous Antiinfective Therapy Due to "Antiinfective Reminders" (AIR Study)
Acronym: AIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FZMI-KEK-ZH-Nr. 2010-0457
Record Dates: First submitted 2011-11-15; First posted 2011-12-26 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Infection as Complication of Medical Care
Keywords: Early reassessment of intravenous antiinfective therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- electronic reminders (Active Comparator): Behavioral: Early switching from intravenous to oral antiinfective agents due to electronic reminders
  Interventions: Other: electronic reminders
- no electronic reminders (No Intervention): Behavioral: Early switching from intravenous to oral antiinfective agents without computerized decision support

INTERVENTIONS:
Other: electronic reminders — Behavioral: Early switching from intravenous to oral antiinfective agents due to electronic reminders
  Other Names: computerized decision support
  Arms: electronic reminders

SUMMARY:
Switching from intravenous application of antiinfective agents to oral therapy is often performed late including high costs and risk of complications. This study will investigate the impact of displayed reminders in the electronic patient chart after 60h of intravenous therapy with an antiinfective agent.

DETAILED DESCRIPTION:
Switching from intravenous application of antiinfective agents to oral therapy is often performed late including high costs, risk of complications as well as higher workload on nursing. This study will investigate the impact of displayed reminders in the electronic patient chart after 60h of intravenous therapy with an antiinfective agent.

ELIGIBILITY:
Inclusion criteria:

* all in-patients in treatment with an intravenous antiinfective for >60h,
* hospitalized in a ward with computerized physician order entry (cpoe)

Exclusion criteria:

* outpatients,
* ward without cpoe,
* no intravenous antiinfective treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74766 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
duration of intravenous antiinfective therapy until switching | 1 year

SECONDARY OUTCOMES:
costs (per year, per day and patient) | 1 year
defined daily doses (per 100 days) | 1 year
duration of hospitalization | 1 year
ratio of narrow to broad-spectrum antibiotics | 1 year
requests for consultations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Blaser, Professor, Principal Investigator — University Hospital Zurich, Center for Clinical Research
Locations (1):
- University Hospital Zurich, Center for Clinical Research, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Beeler PE, Kuster SP, Eschmann E, Weber R, Blaser J. Earlier switching from intravenous to oral antibiotics owing to electronic reminders. Int J Antimicrob Agents. 2015 Oct;46(4):428-33. doi: 10.1016/j.ijantimicag.2015.06.013. Epub 2015 Jul 21. PMID 26293470